CLINICAL TRIAL: NCT00219414
Title: Study for the Treatment of Ulcerative Colitis With Adacolumn (Companion to US Study 512-04-205)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 512-04-205-CS
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Device: Adacolumn Apheresis System

SUMMARY:
The purpose of the study is to demonstrate the safety and effectiveness of the Adacolumn Apheresis System to treat the signs and symptoms of ulcerative colitis.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Treatment, Randomized, Double-Blind, Placebo Control, Parallel Assignment, Safety/Efficacy Study.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 2005-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Primary Outcomes: Effectiveness will be primarily evaluated at Week 12 by disease activity index (DAI) score; Safety will be evaluated by determining the frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lofberg, Prof., Principal Investigator — IBD-unit, Dept. of Gastroenterology, HMQ Sophia Hospital, Stockholm, Sweden; Toshifumi Hibi, Prof., Principal Investigator — Keio University, Tokyo, Japan